CLINICAL TRIAL: NCT05954494
Title: Protection Response to Cellular Stress in BPAN's Patient Study
Acronym: REP-BPAN
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0566
Record Dates: First submitted 2023-07-13; First posted 2023-07-20 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Children and Adults With BPAN Carrying Pathogenic Variants of WDR45
Keywords: BPAN; WDR45; Stress protection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (one sampling of 10 to 20mL for the 4 first patients of the HCL center) which will serve to generate lymphoblastoid cell lines and iPSC (induced pluripotent stem cells - if sampling of 20 mL).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: BPAN Patients — Patients, children or adults with a neurological impairment (epilepsy, dystonia, cognitive impairment...) related to a pathogenic variant of the WDR45 gene

SUMMARY:
BPAN (beta-propeller associated neurodegeneration) is caused by mutations in the autophagy gene WDR45, also known as WIPI4, located on the X chromosome. Mutations in WDR45 result in neurodevelopmental impairment in girls and early-onset epileptic encephalopathy in boys, followed by neurodegeneration in adults (SENDA). This condition is a subtype of neurodegeneration with brain iron overload (NBIA). BPAN is the most recently identified subtype of NBIA and it is important to understand how mutations in WDR45, present in patients∙e∙s, cause cell death.

Autophagy is a cell survival mechanism responsible for the degradation and recycling of cell contents. It has been proposed that autophagy becomes less efficient during normal aging, which could cause neuronal death and thus lead to neurodegeneration.

Reduced autophagic activity has been observed in lymphoblastic cells of BPAN patients and in brains of KO mice for WDR45. The current hypothesis to explain the pathology associated with WDR45 mutations is that a defect in autophagy leads to neurodegeneration. However, we do not know if the autophagy defect is causal or if other deregulations of cellular responses contribute to neurodegeneration. Preliminary results from Pr. Bertrand Mollereau's team suggest that a global deregulation of cellular stress responses may be induced in patient cells. This includes in particular the endoplasmic reticulum response to stress (UPR response) as well as lipid storage mechanisms.

The investigators hypothesize that cells from patients carrying pathogenic variants of WDR45 will exhibit deregulation of cellular stress response pathways.

ELIGIBILITY:
Inclusion Criteria:

* Weight ≥ 12.5kg
* Presence of WDR45 pathogenic variant gene
* Children or adults (no upper limit for age)
* Patient under guardianship could be included if they are assisted by their guardian/adviser in compliance with article L1122-2 of the Public Health Code by virtue of the protection of vulnerable populations

Exclusion Criteria:

- According to the order of 12/04/2018 of the Public Health Code : Weight ≤ 12.5 kg for a 10mL sample or For 2 male and 2 female Lyon patients : Weight ≤ 25 kg for a 20mL sample

* No French Social Insurance Regimen
* Refusal of participation by the legal representative of the patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community sample of patients, organized with patient's associations and major reference centers. As this is a rare genetic disorder with no treatment, we conduct this research at the request of the above-mentioned patient associations.
  At present, about twenty patients are followed for this pathology in France and 2 to 3 patients are diagnosed on average each year. Assuming a refusal rate of 5% (knowing that this study is based on the wishes of the patients' families), we plan to include a total of 20 patients.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-10-23 (Actual); Study Completion 2025-10-23 (Actual)

PRIMARY OUTCOMES:
Autophagic capacity of BPAN cells as marker of cellular stress response | At study completion in an average of 12 months
  * Expression of LC3 protein
  * Expression of p62 protein

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Groupement hospitalier est, Bron, Bron
  - Service de génétique - Laboratoire de Biologie Médicale Multi-Site (LBMMS) Groupement Hospitalier Est - Hospices Civils de Lyon, Bron, Bron

IPD SHARING:
Plan to Share IPD: No